CLINICAL TRIAL: NCT01345370
Title: Comparative Assessment of Methods to Analyze MGMT as a Predictive Factor of Response to Temozolomide in Glioblastomas.
Brief Title: Comparison of Different Methods to Test MGMT Status in Glioblastoma Patients
Acronym: ECOM
Status: Completed | Type: Observational
Sponsor: Center Eugene Marquis (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Veronique QUILLIEN, MD, Center Eugene Marquis
Other Study IDs: ECOM-Glioblastome
Record Dates: First submitted 2011-04-20; First posted 2011-05-02 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Freezed or/and parffine embedded tumor samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stupp protocole: All subjects enrolled must be treated according to the Stupp schedule : surgical resection followed by Temozolomide (TMZ) chemotherapy with concomitant radiotherapy, and then 6 cycles of adjuvant Temzolomide.
  Interventions: Drug: Temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Temozolomide — According to sites procedures
  Other Names: Temodal (brand name).
Radiation: Radiation Therapy — According to sites procedures
  Other Names: Radiotherapy

SUMMARY:
Treatment for newly diagnosed glioblastomas currently involves surgical resection followed by Temozolomide chemotherapy with concomitant radiotherapy, and then 6 cycles of Temozolomide in adjuvant. According to many studies, only those patients not expressing the enzyme repair MGMT benefit from the adjunction of Temozolomide. Therefore, many patients receive unnecessary treatment. The aim of this project is to compare different techniques for analysis of MGMT in order to choose the approach with the best cost/utility ratio, which will allow the selection of patients likely to respond to TMZ chemotherapy during the first course of GBM treatment.

DETAILED DESCRIPTION:
Treatment for newly diagnosed glioblastomas (GBM) currently involves surgical resection followed by Temozolomide (TMZ) chemotherapy with concomitant radiotherapy, and then 6 cycles of TMZ in adjuvant (Stupp schedule). According to many studies, only those patients not expressing the enzyme repair MGMT benefit from the adjunction of TMZ. Therefore, many patients receive unnecessary treatment at an average cost of about 15,000 euros.

The aim of this project is to compare different techniques for analysis of MGMT in order to choose the approach with the best cost/utility ratio, which will allow the selection of patients likely to respond to TMZ chemotherapy during the first course of GBM treatment. Another aspect of this project is to evaluate the extra cost produced by TMZ treatment, and therefore the expected cost saving in the case of using a reliable predictive factor. This kind of evaluation is of great importance, as the MGMT test status is beginning to appear in the decisional care trees of high-grade gliomas The two main techniques for MGMT analysis are currently immunohistochemistry (IH) and molecular analysis of promoter methylation of the gene. Immunohistochemistry is simple and quick, but there is no consensus about labelling or evaluation of the staining, all of which could lead to variability in results. Studies of promoter methylation are currently performed by the MS-PCR technique, in particular the article published in the N Engl J Med in 2005 showing that only patients with a methylated promoter benefit from TMZ adjunction. This technique appears somewhat rudimentary compared to techniques avoiding subjectivity linked to eye reading of the gel after electrophoresis of PCR products.

In phase one of this multicenter national study, IH, MS-PCR, MethyLight, pyrosequencing and MS-HRM will be compared in a retrospective study on 100 samples (frozen for molecular analysis and paraffin-embedded for IH), taken from patients treated according to the Stupp protocol and with a follow-up of 18 months at least. In phase 2, the two techniques with the best cost/efficacy ratio (based on predictive value, analytical quality and feasibility of the test) will be implemented in all the laboratories according to a standard protocol developed by the referral centre for the tests. The dissemination of quality controls will allow us to check that the same results are obtained from one laboratory to another. In phase 3, samples will be analysed prospectively in the different centres and a medico-economic analysis will be undertaken on the integration of MGMT analysis into the standard care of GBM patients. Two types of analysis will be performed: i) on the costs of the techniques, allowing us in particular to estimate the possible additional clinical cost generated and its effect on the cost of a hospital stay, in order to adjust the charging system, and ii) on alternative care strategies for the patients, with or without screening, leading to improve the target of treatments by TMZ, with the aim of improving the definition of "options and recommendations" (cost-utility analysis).

ELIGIBILITY:
Inclusion Criteria:

* Adult, age from 18 to 70
* Pre-surgical diagnosis compatible with a primary or secondary sub-tentorial glioblastoma than can be resected
* No counter-indication to an adjuvant treatment according to the Stupp schedule
* Free written informed consent

Exclusion Criteria:

* Absence of tumor sample available
* Definite histology not related to a glioblastoma or a main oligodendroglioma component

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioblastoma, eligible to resection and to a treatment according to the Stupp schedule.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-03; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Survival of patients according to their MGMT status. | 12 months after last enrollment
  Predictive MGMT methylation tests values related to mean overall survival.

SECONDARY OUTCOMES:
Progression-Free Survival | 12 months

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHRU Hautepierre, Strasbourg, Alsace
  - CHU de Bordeaux, Bordeaux, Aquitaine
  - CHU de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - CHU de Lyon, Lyon, Auvergne-Rhône-Alpes
  - CHU Cote de Nacre, Caen, Basse Normandie
  - Center Eugene Marquis, Rennes, Brittany Region
  - CHRU de Lille, Lille, Hauts-de-France
  - CHU La Timone, Marseille, Paca
  - CHU de Poitiers, Poitiers, Poitou-Charentes
  - CHU La Salpetriere, Paris, Île-de-France Region

REFERENCES:
- [Background] Hegi ME, Diserens AC, Gorlia T, Hamou MF, de Tribolet N, Weller M, Kros JM, Hainfellner JA, Mason W, Mariani L, Bromberg JE, Hau P, Mirimanoff RO, Cairncross JG, Janzer RC, Stupp R. MGMT gene silencing and benefit from temozolomide in glioblastoma. N Engl J Med. 2005 Mar 10;352(10):997-1003. doi: 10.1056/NEJMoa043331. PMID 15758010
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009